CLINICAL TRIAL: NCT00566280
Title: Molecular Breast Imaging: Evaluation of a New Technique Using Scintimammography as an Additional Diagnostic Tool for Women Presenting With a History of Bloody Nipple Discharge and Negative Routine Imaging Studies - A Pilot Study
Brief Title: Molecular Breast Imaging in Patients With a History of Bloody Nipple Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-003072
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer; Bloody Nipple Discharge
Keywords: MBI; Mammogram; Breast Cancer; Breast Ultrasound; Bloody Nipple Discharge; Molecular Breast Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Molecular Breast Imaging (Other)
  Interventions: Procedure: Molecular Breast Imaging

INTERVENTIONS:
Procedure: Molecular Breast Imaging — A dual-detector cadmium-zinc-telluride gamma camera system mounted on a modified mammography gantry is used to image the breast. The injection dose of the radiopharmaceutical given to the patient is 20 mCi of 99m Tc-sestamibi.
  Other Names: MBI

SUMMARY:
The purpose of this study is to evaluate molecular breast imaging in the workup of patients with a history of bloody nipple discharge, not reproducible in the office who have a negative clinical breast examination, and a negative diagnostic mammogram and breast ultrasound.

DETAILED DESCRIPTION:
Although the cause of bloody nipple discharge is benign in most cases, the evaluation is focused on excluding a malignant cause. When bloody nipple discharge is clinically reproducible, management traditionally involves surgical duct excision. When bloody nipple discharge is not reproducible and mammogram and ultrasound are negative the management relies on "watchful waiting" - serial breast imaging to exclude a focal finding and continued observation for recurrent bloody nipple discharge. This approach provokes anxiety among patients who do not have a clear explanation for the bloody nipple discharge. Galactography is useful when positive, but has a high false-negative rate. MRI has not been studied in this context and is costly. Ductoscopy may play a diagnostic role in the future, but experience and equipment are limiting variables. The availability of a less costly method of excluding breast cancer would be of great value in this population.

Molecular Breast Imaging (MBI) is a highly promising novel methodology for breast cancer detection developed under the leadership of Dr. Michael O'Connor at Mayo Clinic, Rochester, MN. Preliminary patient studies with our dual-detector system indicate that this system is capable of reliably detecting very small (5-10 mm) malignant lesions in the breast.

ELIGIBILITY:
Inclusion Criteria:

* Women age 25 - 75
* Women with a negative diagnostic mammogram and ultrasound
* Women with a history of bloody nipple discharge which can not be reproduced by the examining physician or the patient in the office

Exclusion Criteria:

* Pregnant or lactating
* Unable to understand or sign a consent form
* Physically unable to sit upright and still for 40 minutes

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Detection of Breast Cancer | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Wahner-Roedler DL, Hruska CB, O'Connor MK, Phillips SW, Whaley DH, Johnson RE, Degnim AC, Boughey JC, Rhodes DJ. Molecular breast imaging for women presenting with a history of non-reproducible bloody nipple discharge and negative findings on routine imaging studies: a pilot study. J Surg Radiol. 2011 Jan 1;2(3):92-9. Epub 2010 Nov 23.